CLINICAL TRIAL: NCT04338061
Title: A Phase III, Multicenter, Randomized, Parallel Group, Double Blind, Double Dummy, Active Controlled Study of Evobrutinib Compared With Teriflunomide, in Participants With Relapsing Multiple Sclerosis to Evaluate Efficacy and Safety (evolutionRMS 2)
Brief Title: Study of Evobrutinib in Participants With RMS (evolutionRMS 2)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Primary analysis of the RMS phase 3 study (MS200527_0082) resulted in the early termination of the study.
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: EMD Serono Research & Development Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS200527_0082; 2019-004980-36 (EudraCT Number)
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Evobrutinib; Teriflunomide; Aubagio®; Relapsing Multiple Sclerosis
MeSH Terms: interventions — teriflunomide; evobrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Teriflunomide (Active Comparator)
  Interventions: Drug: Teriflunomide
- Evobrutinib (Experimental)
  Interventions: Drug: Evobrutinib

INTERVENTIONS:
Drug: Teriflunomide — Participants received Teriflunomide at a dose of 14 milligrams (mg) orally once daily up to 156 weeks in Double blind treatment period (DBTP) followed by once daily oral doses of Teriflunomide 14 mg up to 96 weeks in double blind extension (DBE) period.
  Arms: Teriflunomide
Drug: Evobrutinib — Participants received Evobrutinib at a dose of 45 mg orally twice daily up to 156 weeks in Double blind treatment period (DBTP) followed by twice daily oral doses of Evobrutinib 45 mg up to 96 weeks in double blind extension (DBE) period.
  Other Names: M2951
  Arms: Evobrutinib

SUMMARY:
The study is to evaluate the efficacy and safety of evobrutinib administered orally twice daily versus Teriflunomide (Aubagio®), administered orally once daily in participants with Relapsing Multiple Sclerosis (RMS). Participants who complete the double-blind treatment period (DBTP) and double-blind extension period (DBEP) prior to approval of a separate long-term follow-up study in their country will get an option for evobrutinib treatment continuation through a 96-week open-label extension (OLE) period.

ELIGIBILITY:
Inclusion Criteria:

* Participants are diagnosed with RMS (relapsing-remitting multiple sclerosis [RRMS] or secondary progressive multiple sclerosis [SPMS] with relapses) in accordance with 2017 Revised McDonald criteria (Thompson 2018)
* Participants with one or more documented relapses within the 2 years before Screening with either: a. one relapse which occurred within the last year prior to randomization, OR b. the presence of at least 1 gadolinium-enhancing (Gd+) T1 lesion within 6 months prior to randomization
* Participants have Expanded Disability Status Scale (EDSS) score of 0 to 5.5 at Screening and Baseline (Day 1). Participants with an EDSS score less than or equal to [<=] 2 at Screening and Baseline (Day 1) are only eligible for participation if their disease duration (time since onset of symptoms) is no more than 10 years
* Participants are neurologically stable for >= 30 days prior to both screening and baseline (Day 1)
* Female participants must be neither pregnant nor breast-feeding or must lack child-bearing potential (as defined by either: post-menopausal or surgically sterile), or use an effective method of contraception for the duration of the study and at least 2 years after study intervention due to the long elimination period for teriflunomide of 2 years, unless the participant undergoes an accelerated elimination procedure
* Male participants must refrain from donating sperm and/or abstain from intercourse with women of child-bearing potential or use an effective method of contraception for the duration of the study and at least 2 years after study intervention due to the long elimination period for teriflunomide of 2 years, unless the participant undergoes an accelerated elimination procedure
* Participants have given written informed consent prior to any study-related procedure
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Participants diagnosed with Progressive MS, in accordance with the 2017 Revised McDonald criteria as follows: a). Participants with Primary Progressive MS. b) Participants with secondary progressive MS without evidence of relapse
* Disease duration more than (>) 10 years in participants with an EDSS =< 2.0 at screening and Baseline (Day 1)
* Immunologic disorder other than MS, or any other condition requiring oral, intravenous (IV), intramuscular, or intra-articular corticosteroid therapy, with the exception of well-controlled Type 2 diabetes mellitus or well controlled thyroid disease
* Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1166 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2024-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (278):
- United States (38):
  - Research Site 752, Cullman, Alabama
  - Research Site 741, Scottsdale, Arizona
  - Research Site 704, Tucson, Arizona
  - Research Site 751, Hanford, California
  - Research Site 737, West Hollywood, California
  - Research Site 759, Colorado Springs, Colorado
  - Research Site 725, Fort Collins, Colorado
  - Research Site 746, Altamonte Springs, Florida
  - Research Site 718, Jacksonville, Florida
  - Research Site 702, Naples, Florida
  - Research Site 740, Orlando, Florida
  - Research Site 726, Port Charlotte, Florida
  - Research Site 719, Sarasota, Florida
  - Research Site 743, Tampa, Florida
  - Research Site 707, Tampa, Florida
  - Research Site 732, Vero Beach, Florida
  - Research Site 705, Weeki Wachee, Florida
  - Research Site 753, West Palm Beach, Florida
  - Research Site 742, Honolulu, Hawaii
  - Research Site 715, Evanston, Illinois
  - Research Site 714, Fort Wayne, Indiana
  - Research Site 744, Lafayette, Indiana
  - Research Site 717, Overland Park, Kansas
  - Research Site 735, Nicholasville, Kentucky
  - Research Site 706, Scarborough, Maine
  - Research Site 738, Detroit, Michigan
  - Research Site 723, St Louis, Missouri
  - Research Site 724, Amherst, New York
  - Research Site 736, Asheville, North Carolina
  - Research Site 712, Chapel Hill, North Carolina
  - Research Site 730, Raleigh, North Carolina
  - Research Site 728, Winston-Salem, North Carolina
  - Research Site 711, Canton, Ohio
  - Research Site 757, Columbus, Ohio
  - Research Site 734, Dayton, Ohio
  - Research Site 748, Philadelphia, Pennsylvania
  - Research Site 703, San Antonio, Texas
  - Research Site 721, Norfolk, Virginia
- Belarus (5):
  - Research Site 143, Grodno
  - Research Site 144, Homyel
  - Research Site 142, Minsk
  - Research Site 141, Vitebsk
  - Research Site 145, Vitebsk
- Brazil (9):
  - Research Site 603, Belo Horizonte
  - Research Site 599, Curitiba
  - Research Site 604, Goiânia
  - Research Site 600, Joinville
  - Research Site 614, Passo Fundo
  - Research Site 591, Porto Alegre
  - Research Site 594, Porto Alegre
  - Research Site 596, Porto Alegre
  - Research Site 609, Vitória
- Bulgaria (16):
  - Research Site 155, Blagoevgrad
  - Research Site 156, Dupnitsa
  - Research Site 157, Pleven
  - Research Site 801, Pleven
  - Research Site 804, Pleven
  - Research Site 805, Plovdiv
  - Research Site 151, Sofia
  - Research Site 152, Sofia
  - Research Site 153, Sofia
  - Research Site 158, Sofia
  - Research Site 159, Sofia
  - Research Site 160, Sofia
  - Research Site 802, Sofia
  - Research Site 803, Sofia
  - Research Site 808, Sofia
  - Research Site 154, Veliko Tarnovo
- Canada (4):
  - Research Site 106, Burnaby
  - Research Site 107, London
  - Research Site 105, Montreal
  - Research Site 101, Ottawa
- France (9):
  - Research Site 455, Bordeaux
  - Research Site 459, Brest
  - Reserach Site 451, Clermont-Ferrand
  - Research Site 458, Limoges
  - Research Site 456, Nîmes
  - Research Site 453, Paris
  - Research Site 457, Pringy
  - Research Site 452, Strasbourg
  - Research Site 454, Tours
- Germany (14):
  - Research Site 172, Augsburg
  - Research Site 177, Berlin
  - Research Site 180, Berlin
  - Research Site 178, Bonn
  - Research Site 179, Cologne
  - Research Site 184, Dresden
  - Research Site 174, Hamburg
  - Research Site 182, Heidelberg
  - Research Site 181, Leipzig
  - Research Site 173, Mainz
  - Research Site 176, Minden
  - Research Site 171, Regensburg
  - Research Site 183, Rostock
  - Research Site 175, Tübingen
- Greece (15):
  - Research Site 194, Athens
  - Research Site 196, Athens
  - Research Site 197, Athens
  - Research Site 201, Athens
  - Research Site 202, Athens
  - Research Site 205, Athens
  - Research Site 207, Athens
  - Reserach Site 206, Athens
  - Research Site 198, Heraklion
  - Research Site 204, Ioannina
  - Research Site 192, Larissa
  - Research Site 199, Marousi
  - Research Site 191, Pátrai
  - Research Site 203, Pátrai
  - Research Site 195, Thessaloniki
- India (4):
  - Research Site 445, Ahmedabad
  - Research Site 444, Bangalore
  - Research Site 443, Mangalore
  - Research Site 442, New Delhi
- Italy (12):
  - Research Site 218, Bari
  - Research Site 216, Catania
  - Research Site 214, Cefalù
  - Research Site 219, Florence
  - Research Site 221, Milan
  - Research Site 211, Napoli
  - Research Site 215, Napoli
  - Research Site 220, Orbassano
  - Research Site 217, Palermo
  - Research Site 212, Pozzilli
  - Research Site 213, Roma
  - Research Site 222, Roma
- Latvia (3):
  - Research Site 231, Riga
  - Research Site 232, Riga
  - Research Site 233, Riga
- Lithuania (4):
  - Research site 241, Kaunas
  - Research site 244, Klaipėda
  - Research site 243, Šiauliai
  - Research site 242, Vilnius
- Malaysia (5):
  - Research Site 551, Kuala Lumpur
  - Research Site 554, Kuala Lumpur
  - Research Site 556, Kuala Lumpur
  - Research Site 552, Kuching
  - Research Site 553, Seberang Jaya
- Moldova (2):
  - Research Site 251, Chisinau
  - Research Site 252, Chisinau
- Norway (3):
  - Research Site 481, Bergen
  - Research site 483, Drammen
  - Research Site 482, Namsos
- Philippines (2):
  - Research Site 562, Baguio City
  - Research Site 561, Cebu City
- Poland (19):
  - Reserach Site 267, Bydgoszcz
  - Reserach Site 268, Bydgoszcz
  - Research Site 273, Katowice
  - Research site 846, Katowice
  - Research site 274, Katowice-Ochojec
  - Research Site 276, Krakow
  - Research Site 263, Lodz
  - Research Site 272, Lodz
  - Research Site 266, Nowa Sól
  - Research Site 270, Poznan
  - Research Site 262, Rzeszów
  - Research Site 265, Siemianowice Śląskie
  - Research Site 271, Szczecin
  - Research Site 264, Warsaw
  - Research Site 277, Warsaw
  - Reserach Site 275, Warsaw
  - Research Site 269, Wroclaw
  - Research Site 261, Zabrze
  - Research Site 278, Zamość
- Portugal (11):
  - Research Site 293, Aveiro
  - Research Site 282, Braga
  - Research Site 289, Coimbra
  - Research Site 281, Lisbon
  - Research Site 283, Lisbon
  - Research Site 287, Lisbon
  - Research SIte 284, Matosinhos Municipality
  - Research Site 292, Porto
  - Research Site 288, Pragal
  - Research Site 291, Santa Maria da Feira
  - Research Site 286, Torres Vedras
- Research Site 791, Guaynabo, Puerto Rico
- Romania (4):
  - Research Site 314, Brasov
  - Research Site 307, Bucharest
  - Research Site 309, Caracal
  - Research Site 302, Târgu Mureş
- Russia (23):
  - Research Site 325, Kazan'
  - Research Site 329, Kazan'
  - Research Site 323, Kemerovo
  - Research Site 344, Kirov
  - Research Site 340, Krasnodar
  - Research Site 334, Krasnoyarsk
  - Research Site 341, Moscow
  - Research Site 343, Moscow
  - Research Site 345, Moscow
  - Research Site 332, Nizhny Novgorod
  - Research Site 327, Novosibirsk
  - Research Site 330, Novosibirsk
  - Research Site 331, Novosibirsk
  - Research Site 335, Novosibirsk
  - Research Site 328, Rostov-on-Don
  - Research Site 324, Saint Petersburg
  - Research Site 338, Saint Petersburg
  - Research Site 339, Saint Petersburg
  - Research Site 342, Saint Petersburg
  - Research Site 346, Saint Petersburg
  - Research Site 326, Saransk
  - Research Site 321, Sestroretsk
  - Research Site 337, Tyumen
- Research Site 493, Riyadh, Saudi Arabia
- Singapore (2):
  - Research Site 571, Singapore
  - Research site 572, Singapore
- Slovakia (8):
  - Research Site 351, Banská Bystrica
  - Research Site 352, Bratislava
  - Research Site 353, Bratislava
  - Research Site 354, Bratislava
  - Research Site 356, Bratislava
  - Research Site 359, Dubnica nad Váhom
  - Research Site 358, Trenčín
  - Research Site 357, Trnava
- Slovenia (3):
  - Research Site 373, Celje
  - Research Site 372, Ljubljana
  - Research Site 371, Maribor
- South Africa (4):
  - Research Site 501, Cape Town
  - Research Site 502, Cape Town
  - Research Site 503, Cape Town
  - Research Site 504, Pretoria
- Spain (12):
  - Research Site 384, Alcorcón
  - Research Site 391, Barakaldo
  - Research Site 390, Barcelona
  - Research Site 382, Córdoba
  - Research Site 389, El Palmar
  - Research Site 388, Madrid
  - Research Site 392, Majadahonda
  - Research Site 383, Málaga
  - Research Site 387, Seville
  - Research Site 385, Valencia
  - Research Site 386, Valencia
  - Research Site 381, Vigo
- Sweden (4):
  - Research Site 512, Gothenburg
  - Research site 514, Malmo
  - Research Site 511, Stockholm
  - Research Site 513, Uppsala
- Switzerland (3):
  - Research Site 404, Aarau
  - Research Site 402, Bern
  - Research Site 403, Lugano
- Thailand (2):
  - Research Site 583, Bangkoknoi
  - Research Site 582, Muang
- Turkey (Türkiye) (13):
  - Research Site 538, Ankara
  - Research Site 544, Ankara
  - Research Site 531, Istanbul
  - Research Site 534, Istanbul
  - Research Site 536, Istanbul
  - Research Site 541, Istanbul
  - Research Site 543, Istanbul
  - Research Site 539, Izmir
  - Research Site 533, Kocaeli
  - Research Site 537, Konya
  - Research Site 540, Mersin
  - Research Site 535, Samsun
  - Research Site 532, Trabzon
- Ukraine (23):
  - Research Site 415, Chernihiv
  - Research Site 417, Chernihiv
  - Research Site 414, Dnipro
  - Research Site 416, Dnipro
  - Research Site 420, Dnipro
  - Research Site 413, Ivano-Frankivsk
  - Research Site 624, Kharkiv
  - Research Site 632, Kharkiv
  - Research Site 633, Kharkiv
  - Research Site 419, Kherson
  - Research Site 411, Kyiv
  - Research Site 418, Kyiv
  - Research Site 629, Lutsk
  - Research Site 627, Lviv
  - Research Site 622, Poltava
  - Research Site 625, Rivne
  - Research Site 628, Ternopil
  - Research Site 630, Uzhhorod
  - Research Site 623, Vinnytsia
  - Research Site 412, Zaporizhzhia
  - Research Site 621, Zaporizhzhia
  - Research Site 631, Zaporizhzhia
  - Research Site 626, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Result] Montalban X, Vermersch P, Arnold DL, Bar-Or A, Cree BAC, Cross AH, Kubala Havrdova E, Kappos L, Stuve O, Wiendl H, Wolinsky JS, Dahlke F, Le Bolay C, Shen Loo L, Gopalakrishnan S, Hyvert Y, Javor A, Guehring H, Tenenbaum N, Tomic D; evolutionRMS investigators. Safety and efficacy of evobrutinib in relapsing multiple sclerosis (evolutionRMS1 and evolutionRMS2): two multicentre, randomised, double-blind, active-controlled, phase 3 trials. Lancet Neurol. 2024 Nov;23(11):1119-1132. doi: 10.1016/S1474-4422(24)00328-4. Epub 2024 Sep 19. PMID 39307151
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527_0082
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Period: Double-blind Treatment Period: 156 Weeks
Arm/Group | Teriflunomide | Evobrutinib
Started | 583 | 583
Completed | 409 | 410
Not Completed | 174 | 173
Not completed — Withdrawal by Subject | 59 | 52
Not completed — Lack of Efficacy | 11 | 16
Not completed — Other Reasons | 17 | 22
Not completed — Adverse Event | 67 | 70
Not completed — Protocol Non-Compliance | 9 | 8
Not completed — Lost to Follow-up | 11 | 3
Not completed — Randomized, but not treated | 0 | 2
Period: Double-blind Extension Period: 96 Weeks
Arm/Group | Teriflunomide | Evobrutinib
Started | 390 | 389
Completed | 381 | 377
Not Completed | 9 | 12
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Non-Compliance | 1 | 0
Not completed — Other Reasons | 4 | 8

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriflunomide | Evobrutinib | Total
Number analyzed (Participants) | 583 | 583 | 1166
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37 (9.5) | 36 (9.1) | 37 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 370 | 413 | 783
  Male | 213 | 170 | 383
Race/Ethnicity, Customized [Number; unit: Participants]
  Ethnicity-Hispanic or Latino | 30 | 51 | 81
  Ethnicity-Not Hispanic or Latino | 553 | 531 | 1084
  Ethnicity-Unknown or Not Reported | 0 | 1 | 1
  Race-American Indian or Alaska Native | 1 | 1 | 2
  Race-Asian | 17 | 15 | 32
  Race-Black or African American | 4 | 4 | 8
  Race-Multiple | 7 | 2 | 9
  Race-Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Race-Other | 1 | 2 | 3
  Race-Unknown or Not Reported | 2 | 2 | 4
  Race-White | 551 | 556 | 1107

OUTCOME MEASURES:

1. Primary Outcome: Double Blind Treatment Period (DBTP) and Double Blind Extension (DBE) Period: Annualized Relapse Rate (ARR)
Description: The qualifying relapse is the occurrence of new or worsening neurological symptoms attributable to Multiple Sclerosis (MS) (for more than [>] 24 hours, no fever, infection, injury, adverse events (AEs), and preceded by a stable or improving neurological state for more than or equal to [>=] 30 days).
Time Frame: Baseline up to 170 weeks
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment.
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 583 | 583
relapses per year | 0.11 [0.09 to 0.13] | 0.11 [0.09 to 0.13]

2. Secondary Outcome: DBTP and DBE Period: Percentage of Participants Without 12-Week Confirmed Disability Progression (CDP) as Measured by Expanded Disability Status Scale (EDSS)
Description: Disability progression was defined as increase in EDSS of greater than or equal to [>=] 1 point from baseline EDSS score, if EDSS score at baseline is 5.0 or less and an increase of >=0.5 point, if the baseline score is 5.5. Disability progression is considered sustained for 12 weeks when the initial increase in the EDSS is confirmed at a regularly scheduled visit at least 12 weeks after the initial documentation of neurological worsening. The total EDSS score ranges from 0 (normal) to 10 (death due to multiple sclerosis). Kaplan-Meier method was used to estimate the percentage of participants without 12-week CDP.
Time Frame: Week 96 and Week 156 (combined DBTP and DBE periods)
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment. The result reported for this outcome measure are the results from data of combined DBTP and DBE periods.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 583 | 583
percentage of participants
  Week 96 | 88.9 [85.7 to 91.4] | 91.8 [88.9 to 93.9]
  Week 156 | 82.3 [76.0 to 87.1] | 85.0 [77.8 to 90.0]

3. Secondary Outcome: DBTP and DBE Period: Percentage of Participants Without 24-Week Confirmed Disability Progression (CDP) as Measured by Expanded Disability Status Scale (EDSS)
Description: Disability progression was defined as increase in EDSS of greater than or equal to [>=] 1 point from baseline EDSS score, if EDSS score at baseline is 5.0 or less and an increase of >=0.5 point, if the baseline score is 5.5. Disability progression is considered sustained for 24 weeks when the initial increase in the EDSS is confirmed at a regularly scheduled visit at least 24 weeks after the initial documentation of neurological worsening. The total EDSS score ranges from 0 (normal) to 10 (death due to multiple sclerosis). Kaplan-Meier method was used to estimate the percentage of participants without 24-week CDP.
Time Frame: Week 96 and Week 156 (combined DBTP and DBE periods)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 583 | 583
percentage of participants
  Week 96 | 91.6 [88.7 to 93.8] | 93.6 [91.0 to 95.5]
  Week 156 | 89.7 [86.5 to 92.2] | 90.9 [87.8 to 93.3]

4. Secondary Outcome: DBTP and DBE Period: Percentage of Participants With 24-Week Confirmed Disability Improvement (CDI) as Measured by Expanded Disability Status Scale (EDSS)
Description: Disability improvement was defined as a reduction of 1 point from Baseline EDSS score when the Baseline score is >= 2 and less than or equal to [<=] 6 and a reduction of 0.5 point from Baseline EDSS score when the Baseline score is >= 6.5 and <= 9.5. Disability improvement is considered sustained when the initial reduction in the EDSS score is confirmed at a regularly scheduled visit at least 24 weeks after the initial reduction. The total EDSS score ranges from 0 (normal) to 10 (death due to multiple sclerosis). Kaplan-Meier method was used to estimate the percentage of participants with 12-week CDI.
Time Frame: Week 96 and Week 156 (combined DBTP and DBE periods)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 583 | 583
percentage of participants
  Week 96 | 11.4 [8.6 to 15.0] | 7.6 [5.4 to 10.7]
  Week 156 | 12.5 [9.5 to 16.4] | 8.4 [6.0 to 11.6]

5. Secondary Outcome: DBTP and DBE Period: Change From Baseline in Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) Score at Week 48, Week 96, Week 120, Week 144 and Week 156
Description: Physical function was assessed with PROMISnq Short Form v2.0 - Physical Function - Multiple Sclerosis 15a (PROMISnq PF(MS) 15a). PROMISnq PF(MS) 15a assesses a participant's abilities and limitations with respect to everyday physical activities. Results are reported as a T-score. In the general population, T-scores have a mean of 50, standard deviation of 10, and range from 10 to 65. Higher T-scores represent higher physical function. Change from baseline in PROMIS PF score was analyzed using Mixed Effect Model for Repeated Measures (MMRM) to evaluate the result of the 2 periods (DBTP and DBE).
Time Frame: Baseline, Week 48, Week 96, Week 120, Week 144 and Week 156 (Combined DBTP and DBE periods)
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment. Here, Overall number of participants analyzed signifies those participants who were evaluable for this outcome measure. The result reported for this outcome measure are the results from data of combined DBTP and DBE periods.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 572 | 572
units on a scale
  Week 48 | 0.25 [-0.22 to 0.72] | 0.31 [-0.16 to 0.78]
  Week 96 | -0.31 [-0.88 to 0.26] | -0.45 [-1.03 to 0.13]
  Week 120 | -0.56 [-1.23 to 0.11] | -0.19 [-0.86 to 0.48]
  Week 144 | -0.38 [-1.12 to 0.35] | -0.57 [-1.31 to 0.17]
  Week 156 | NA [NA to NA] — Week 156 is not evaluable in the modelling due to the lack of participants in some of the covariate categories at that visit. | NA [NA to NA] — Week 156 is not evaluable in the modelling due to the lack of participants in some of the covariate categories at that visit.

6. Secondary Outcome: DBTP and DBE Period: Change From Baseline in Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Score at Week 48, Week 96, Week 120, Week 144 and Week 156
Description: PROMIS Fatigue score was assessed with PROMIS Short Form v1.0 - Fatigue - Multiple Sclerosis 8a (PROMIS Fatigue (MS) 8a). PROMIS Fatigue (MS) 8a assesses level of fatigue and its interference on daily activities. Results are reported as a T-score. In the general population, T-scores have a mean of 50, standard deviation of 10, and range from 33 to 85. Higher T-scores represent higher fatigue. Change from baseline in PROMIS fatigue score was analyzed using Mixed Effect Model for Repeated Measures (MMRM) to evaluate the result of the 2 periods (DBTP and DBE).
Time Frame: Baseline, Week 48, Week 96, Week 120, Week 144 and Week 156 ((combined DBTP and DBE periods)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 572 | 572
units on a scale
  Week 48 | -2.20 [-2.81 to -1.60] | -2.59 [-3.19 to -1.98]
  Week 96 | -2.17 [-2.85 to -1.49] | -2.12 [-2.81 to -1.44]
  Week 120 | -2.24 [-3.00 to -1.48] | -2.59 [-3.35 to -1.83]
  Week 144 | -2.41 [-3.35 to -1.48] | -2.16 [-3.10 to -1.22]
  Week 156 | -2.21 [-3.62 to -0.81] | -2.34 [-3.83 to -0.86]

7. Secondary Outcome: DBTP and DBE Period: Total Number of T1 Gadolinium-positive (Gd+) Lesions
Description: Analysis of Gadolinium-positive T1 lesions was done using magnetic resonance imaging (MRI) scans.
Time Frame: Baseline up to 170 weeks
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment. Here, Overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: lesions per scan
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 544 | 544
lesions per scan | 0.29 [0.24 to 0.34] | 0.51 [0.43 to 0.60]

8. Secondary Outcome: DBTP and DBE Period: New or Enlarging T2 Lesions Rate
Description: Analysis of new or enlarging T2 lesions rate was done using magnetic resonance imaging (MRI) scans. Negative binomial model for lesion count (summed over scans) includes treatment and covariates based on randomization strata and baseline volume of T2 lesion (continuous), with offset equal to the log of the time in years between the last available MRI scan and the baseline scan.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: lesions per year
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 544 | 544
lesions per year | 6.88 [6.01 to 7.87] | 6.17 [5.38 to 7.07]

9. Secondary Outcome: DBTP Period: Neurofilament Light Chain (NfL) Concentration at Week 12
Description: NfL is a biomarker of neuro-axonal damage whose concentration was assessed in blood at Week 12.
Time Frame: Week 12
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram per liter (ng/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 544 | 544
nanogram per liter (ng/L) | 13.09 [12.69 to 13.50] | 12.51 [12.13 to 12.90]

10. Secondary Outcome: DBTP and DBE Periods: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Adverse Events of Special Interest (AESIs)
Description: Adverse event (AE): Any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the study drug. Serious AE: an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs: those AEs with an onset date on or after the date of first study intervention administration, or AEs present prior to any study intervention administration but exacerbating after. TEAEs included both Serious TEAEs and non-serious TEAEs. AESIs included liver AEs (possible drug-induced, non-infectious, non-alcoholic, and immune-mediated), infections (serious and opportunistic infections), lipase and amylase elevation, and seizure.
Time Frame: Baseline up to 170 weeks
Population: Safety (SAF) analysis set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 583 | 581
Participants
  Participants with TEAEs | 524 | 508
  Participants with AESIs | 144 | 135

11. Secondary Outcome: DBTP and DBE Periods: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Severity
Description: Severity of adverse events (AE) were assessed by the investigator per the National Cancer Institute- Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0. Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Death. Number of participants with Grades 1, 2, 3, 4 and 5 were reported.
Time Frame: Baseline up to 170 weeks
Population: Safety (SAF) analysis set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 583 | 581
Participants
  Participants with Grade 1 | 41 | 59
  Participants with Grade 2 | 389 | 351
  Participants with Grade 3 | 87 | 92
  Participants with Grade 4 | 7 | 6
  Participants with Grade 5 | 0 | 0

12. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Vital Signs: Diastolic Blood Pressure and Systolic Blood Pressure
Description: Diastolic blood pressure and systolic blood pressure were measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Changes in vital signs: diastolic blood pressure and systolic blood pressure from baseline up to 170 weeks were reported.
Time Frame: Baseline up to 170 weeks
Population: Safety (SAF) analysis set included all participants who received at least one dose of study treatment. Here, Overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 457 | 454
millimeter of mercury (mmHg)
  Systolic Blood Pressure | 2.4 (11.0) | 1.0 (11.50)
  Diastolic Blood Pressure | 1.4 (8.73) | -0.5 (8.38)

13. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Vital Signs: Pulse Rate
Description: Pulse rate was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Changes in vital signs: pulse rate from baseline up to 170 weeks was reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 457 | 454
beats per minute | 2.2 (10.19) | 3.0 (10.15)

14. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Vital Signs: Respiratory Rate
Description: Respiratory rate was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Changes in vital signs: respiratory rate from baseline up to 170 weeks was reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 457 | 454
breaths per minute | -0.3 (1.75) | -0.5 (1.87)

15. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Vital Signs: Weight
Description: Changes in vital signs: weight from baseline up to 170 weeks was reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 457 | 454
kilograms (kg) | -0.51 (5.447) | 1.06 (5.310)

16. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Vital Signs: Temperature
Description: Temperature was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Changes in vital signs: Temperature from baseline up to 170 weeks was reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 457 | 454
degree Celsius | -0.02 (0.340) | -0.03 (0.350)

17. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Electrocardiograms (ECGs): Heart Rate
Description: Heart rate was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Changes in vital signs: heart rate from baseline up to 170 weeks was reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 77 | 69
beats per minute | -0.1 (10.36) | 2.6 (10.20)

18. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Electrocardiograms (ECGs): QT Interval - Fridericia's Correction Formula, PR Interval and QRS Duration
Description: QT Interval - Fridericia's Correction Formula, PR Interval and QRS Duration was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Changes in vital signs: QT Interval - Fridericia's Correction Formula, PR Interval and QRS Duration from baseline up to 170 weeks were reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 77 | 69
milliseconds (msec)
  QT Interval - Fridericia's Correction Formula | -2.14 (16.459) | -0.07 (14.935)
  PR Interval | -4.2 (16.82) | -3.1 (14.51)
  QRS Duration | -2.8 (6.77) | -1.1 (8.94)

19. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Hematology Parameter: Hemoglobin and Erythrocytes Mean Corpuscular Hemoglobin (HGB) Concentration
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameters: erythrocytes mean corpuscular HGB concentration and hemoglobin. Changes in hematology parameters: erythrocytes mean corpuscular HGB concentration and hemoglobin from baseline up to 170 weeks were reported.
Time Frame: Baseline up to 170 weeks
Population: Safety (SAF) analysis set included all participants who received at least one dose of study treatment. Here, Overall number of participants analyzed signifies those participants who were evaluable for this outcome measure and "number analyzed"= participants who were evaluable for the specified categories.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 447 | 436
gram per liter (g/L)
  Erythrocytes Mean Corpuscular HGB Concentration: number analyzed (Participants) | 438 | 428
  Erythrocytes Mean Corpuscular HGB Concentration | 0.0 (11.07) | -1.9 (12.42)
  Hemoglobin | -3.4 (11.40) | -3.4 (11.43)

20. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Hematology Parameter: Platelets, Leukocytes, Neutrophils, Eosinophils, Basophils, Monocytes, Lymphocytes and Reticulocytes
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameters: Platelets, Leukocytes, Neutrophils, Eosinophils, Basophils, Monocytes, Lymphocytes and Reticulocytes. Changes in hematology parameters: Platelets, Leukocytes, Neutrophils, Eosinophils, Basophils, Monocytes, Lymphocytes and Reticulocytes from baseline up to 170 weeks were reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 446 | 437
10^9 cells per liter
  Platelets: number analyzed (Participants) | 441 | 432
  Platelets | -8.4 (48.38) | 9.8 (52.24)
  Leukocytes | -0.39 (1.954) | 0.24 (1.883)
  Neutrophils: number analyzed (Participants) | 331 | 324
  Neutrophils | -0.471 (1.7550) | 0.156 (1.7796)
  Eosinophils: number analyzed (Participants) | 438 | 431
  Eosinophils | 0.0198 (0.14809) | 0.0238 (0.14945)
  Basophils: number analyzed (Participants) | 438 | 431
  Basophils | -0.0081 (0.03882) | -0.0042 (0.03902)
  Monocytes: number analyzed (Participants) | 438 | 432
  Monocytes | 0.0797 (0.19710) | 0.0772 (0.20715)
  Lymphocytes: number analyzed (Participants) | 442 | 434
  Lymphocytes | -0.0241 (0.57564) | 0.0311 (0.57810)
  Reticulocytes: number analyzed (Participants) | 436 | 430
  Reticulocytes | 2.001 (23.3886) | -0.841 (20.2200)

21. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Hematology Parameters: Hematocrit
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameter: Hematocrit. Changes in hematology parameter: Hematocrit from baseline up to 170 weeks was reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 442 | 431
percentage of cells | -0.0107 (0.03199) | -0.0085 (0.03311)

22. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameter: Erythrocytes Mean Corpuscular Hemoglobin. Changes in hematology parameter: Erythrocytes Mean Corpuscular Hemoglobin from baseline up to 170 weeks was reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: picogram
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 443 | 435
picogram | -0.44 (1.603) | -0.93 (1.941)

23. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameter: Erythrocytes Mean Corpuscular Volume. Changes in hematology parameter: Erythrocytes Mean Corpuscular Volume from baseline up to 170 weeks was reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 441 | 431
femtoliters | -1.48 (4.150) | -2.53 (5.217)

24. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Biochemistry Parameters: Bilirubin and Creatinine
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the biochemistry parameters: Bilirubin and Creatinine. Changes in biochemistry parameters: Bilirubin and Creatinine from baseline up to 170 weeks were reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: micromoles per liter (mcmol/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 455 | 446
micromoles per liter (mcmol/L)
  Bilirubin | -0.02 (4.649) | 0.33 (4.212)
  Creatinine: number analyzed (Participants) | 449 | 442
  Creatinine | 1.6 (8.93) | 2.4 (12.06)

25. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Biochemistry Parameters: Aspartate Aminotransferase, Alanine Aminotransferase, Alkaline Phosphatase, Amylase, Lipase, Gamma Glutamyl Transferase and Lactate Dehydrogenase
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the biochemistry parameters: Aspartate Aminotransferase, Alanine Aminotransferase, Alkaline Phosphatase, Amylase, Lipase, Gamma Glutamyl Transferase and Lactate Dehydrogenase. Changes in biochemistry parameters: Aspartate Aminotransferase, Alanine Aminotransferase, Alkaline Phosphatase, Amylase, Lipase, Gamma Glutamyl Transferase and Lactate Dehydrogenase from baseline up to 170 weeks were reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 455 | 446
units per liter (U/L)
  Aspartate Aminotransferase: number analyzed (Participants) | 454 | 444
  Aspartate Aminotransferase | 2.64 (15.365) | 1.74 (13.219)
  Alanine Aminotransferase | 4.40 (33.878) | 2.75 (32.018)
  Alkaline Phosphatase: number analyzed (Participants) | 447 | 445
  Alkaline Phosphatase | 2.32 (15.875) | 6.69 (15.659)
  Amylase: number analyzed (Participants) | 450 | 441
  Amylase | 1.3 (14.42) | 2.1 (15.91)
  Lipase: number analyzed (Participants) | 449 | 442
  Lipase | -0.3 (18.35) | 2.3 (17.26)
  Gamma Glutamyl Transferase: number analyzed (Participants) | 359 | 385
  Gamma Glutamyl Transferase | 3.71 (26.084) | 1.98 (20.207)
  Lactate Dehydrogenase: number analyzed (Participants) | 436 | 439
  Lactate Dehydrogenase | 7.08 (27.049) | -5.41 (27.637)

26. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Biochemistry Parameters: Sodium, Potassium, Calcium, Magnesium, Glucose, Chloride, Urea Nitrogen, Phosphate, Bicarbonate and Corrected Calcium
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the biochemistry parameters: Sodium, Potassium, Calcium, Magnesium, Glucose, Chloride, Urea Nitrogen, Phosphate, Bicarbonate and Corrected Calcium. Changes in biochemistry parameters: Sodium, Potassium, Calcium, Magnesium, Glucose, Chloride, Urea Nitrogen, Phosphate, Bicarbonate and Corrected Calcium from baseline up to 170 weeks were reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 450 | 446
millimole per liter (mmol/L)
  Sodium: number analyzed (Participants) | 448 | 440
  Sodium | 0.9286 (2.56796) | 0.7750 (3.21185)
  Potassium: number analyzed (Participants) | 449 | 439
  Potassium | 0.0405 (0.48750) | 0.0376 (0.44331)
  Calcium: number analyzed (Participants) | 448 | 440
  Calcium | -0.006 (0.1197) | -0.008 (0.1121)
  Magnesium: number analyzed (Participants) | 449 | 441
  Magnesium | -0.002 (0.0656) | -0.006 (0.0667)
  Glucose: number analyzed (Participants) | 448 | 440
  Glucose | 0.09 (0.949) | 0.16 (0.812)
  Chloride: number analyzed (Participants) | 450 | 440
  Chloride | 2.3 (3.30) | 2.1 (3.53)
  Urea Nitrogen: number analyzed (Participants) | 447 | 441
  Urea Nitrogen | 0.126 (1.2759) | 0.122 (1.1651)
  Phosphate: number analyzed (Participants) | 428 | 434
  Phosphate | -0.047 (0.1944) | -0.024 (0.1799)
  Bicarbonate: number analyzed (Participants) | 324 | 348
  Bicarbonate | 0.44 (2.592) | 0.17 (2.980)
  Corrected Calcium: number analyzed (Participants) | 446 | 437
  Corrected Calcium | 0.0290 (0.10405) | 0.0292 (0.09775)

27. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Biochemistry Parameters: Total Protein and Albumin
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the biochemistry parameters: Total Protein and Albumin. Changes in biochemistry parameters: Total Protein and Albumin from baseline up to 170 weeks were reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 448 | 444
gram per liter (g/L)
  Total protein: number analyzed (Participants) | 448 | 437
  Total protein | -1.31 (4.905) | -0.59 (4.998)
  Albumin | -1.75 (3.497) | -1.83 (3.287)

28. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Biochemistry Parameters: Glomerular Filtration Rate
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the biochemistry parameter: Glomerular Filtration Rate. Changes in biochemistry parameter: Glomerular Filtration Rate from baseline up to 170 weeks were reported. The Glomerular Filtration Rate was measured as milliliter per minute per 1.73 square meter (mL/min/1.73m^2).
Time Frame: Baseline up to 170 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 360 | 351
mL/min/1.73m^2 | -4.7 (13.41) | -5.7 (13.81)

29. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Urinalyses Parameter: Potential of Hydrogen (pH) of Urine
Description: Urine samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the urinalyses parameter: pH. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Changes in urinalyses parameter: pH from baseline up to 170 weeks was reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 442 | 438
pH | -0.03 (0.936) | -0.04 (0.973)

30. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Urinalyses Parameter: Specific Gravity of Urine
Description: Urine samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the urinalyses parameter: Specific Gravity of Urine. Changes in urinalyses parameter: Specific Gravity of Urine from baseline up to 170 weeks was reported.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Kilogram per cubic meter
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 436 | 428
Kilogram per cubic meter | -0.0015 (0.04460) | -0.0017 (0.03748)

31. Secondary Outcome: DBTP and DBE Periods: Absolute Concentrations of Immunoglobulin (Ig) Levels
Description: Absolute Concentrations serum levels of IgG, IgA, IgM were assessed.
Time Frame: At Week 170
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 319 | 341
gram per liter (g/L)
  IgA | 1.899 (0.7787) | 2.581 (1.1201)
  IgG | 10.082 (2.1551) | 10.990 (2.4844)
  IgM | 1.251 (0.6445) | 1.196 (0.6151)

32. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Immunoglobulin (Ig) Levels
Description: Change from baseline serum levels of IgG, IgA, IgM were assessed.
Time Frame: Baseline up to 170 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 319 | 339
gram per liter (g/L)
  IgA | -0.203 (0.5704) | 0.500 (0.7197)
  IgG | -0.645 (1.6188) | 0.146 (1.8712)
  IgM | -0.167 (0.5094) | -0.175 (0.3888)

ADVERSE EVENTS:
Time Frame: Baseline up to 170 weeks
Description: Safety (SAF) analysis set included all participants who received at least one dose of study treatment.
Arm/Group | Teriflunomide | Evobrutinib
All-Cause Mortality (participants affected / at risk) | 0/583 | 0/581
Serious Adverse Events (participants affected / at risk) | 37/583 | 51/581
Other Adverse Events (participants affected / at risk) | 455/583 | 409/581
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriflunomide (N=583) | Evobrutinib (N=581)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 1 (1)
Ileus spastic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Salpingo-oophoritis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bladder injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary tract injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (3)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Symphysiolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Synovial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Autonomic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 1 (2) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1) | 3 (3)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1)
Neuropsychiatric symptoms (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Miscarriage of partner (Social circumstances) | 0 (0) | 1 (1)
Pregnancy of partner (Social circumstances) | 0 (0) | 1 (1)
Subgaleal haematoma (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriflunomide (N=583) | Evobrutinib (N=581)
Anaemia (Blood and lymphatic system disorders) | 23 (35) | 34 (54)
Neutropenia (Blood and lymphatic system disorders) | 47 (112) | 22 (33)
Diarrhoea (Gastrointestinal disorders) | 47 (59) | 24 (28)
Nausea (Gastrointestinal disorders) | 36 (39) | 29 (39)
Fatigue (General disorders) | 47 (66) | 37 (46)
COVID-19 (Infections and infestations) | 121 (139) | 105 (119)
Nasopharyngitis (Infections and infestations) | 67 (103) | 58 (89)
Respiratory tract infection viral (Infections and infestations) | 37 (52) | 23 (36)
Upper respiratory tract infection (Infections and infestations) | 45 (81) | 55 (83)
Urinary tract infection (Infections and infestations) | 33 (46) | 39 (49)
Alanine aminotransferase increased (Investigations) | 126 (227) | 99 (168)
Aspartate aminotransferase increased (Investigations) | 80 (123) | 61 (84)
Gamma-glutamyltransferase increased (Investigations) | 29 (70) | 31 (37)
Lipase increased (Investigations) | 33 (39) | 33 (55)
Lymphocyte count decreased (Investigations) | 39 (73) | 27 (40)
Neutrophil count decreased (Investigations) | 92 (156) | 40 (42)
White blood cell count decreased (Investigations) | 63 (122) | 23 (39)
Back pain (Musculoskeletal and connective tissue disorders) | 61 (79) | 49 (63)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 32 (40) | 30 (46)
Headache (Nervous system disorders) | 103 (169) | 96 (198)
Alopecia (Skin and subcutaneous tissue disorders) | 84 (87) | 35 (38)

LIMITATIONS AND CAVEATS:
The Final Analysis represents the analysis of the cumulative data collected up to the Primary Analysis trigger and beyond through DBE up to the final database lock. Therefore, the endpoints were evaluated considering a time period from the start of DBTP to the end of the DBE Period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT04338061/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT04338061/SAP_001.pdf